CLINICAL TRIAL: NCT06434194
Title: Serranator OCT: Understanding the Mechanism of Action of Serration Angioplasty by Serranator Versus Conventional Balloon Angioplasty for below-the Knee (BTK) Artery Disease Using Optical Coherence Tomography (OCT)
Brief Title: Serrantor OCT Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cagent Vascular LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSP
Record Dates: First submitted 2024-05-03; First posted 2024-05-30 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Critical Limb Ischemia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Serrantor (Active Comparator): Subjects randomized to the Serranator Arm of the study will be treated with the Serranator PTA Serration Balloon
  Interventions: Device: Serranator PTA Serration Catheter
- PTA (Active Comparator): Subjects randomized to the PTA Arm of the study will be treated with a standard of care percutaneous transluminal angioplasty (PTA) balloon.
  Interventions: Drug: PTA (Standard of Care)

INTERVENTIONS:
Device: Serranator PTA Serration Catheter — The Serranator PTA Serration Balloon Catheter is an over-the-wire balloon dilatation catheter designed to perform percutaneous transluminal angioplasty (PTA) for peripheral indications.
  Arms: Serrantor
Drug: PTA (Standard of Care) — A percutaneous transluminal angioplasty catheter will be used to treat the target lesion.
  Arms: PTA

SUMMARY:
TA prospective randomized control trial to evaluate the serration angioplasty effect in BTK arteries with varying degrees of calcified plaque.

ELIGIBILITY:
Inclusion Criteria:

* Rutherford clinical category 4-6 of the target limb
* Age of subjects is >18 years old
* Patients has given informed consent to participate in this study

Exclusion Criteria:

* De novo or restenotic (without prior stent) stenosis (≥70%) or occlusion
* Target lesion is in the BTK arteries, including below the knee popliteal, tibioperoneal trunk, tibial, peroneal, and pedal arteries.
* Angiographic visual estimated reference vessel diameter is between 2.0 and 5.0 mm.
* Lesion length less than 220 mm

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Residual Lumen Volume Stenosis | Baseline
  Residual lumen volume stenosis derived by OCT comparing Serration Angioplasty and conventional plain balloon angioplasty (PTA) measured at 10-15min post procedure. The lesion segment is defined as the entire treated segment where the balloon has been inflated.

SECONDARY OUTCOMES:
OCT Residual Diameter Stenosis | Baseline
  Residual stenosis as measured by OCT
Angiography Residual Diameter Stenosis | Baseline
  Residual stenosis as measured by angiography
Dissection Pattern | Baseline
  The incidence of dissection pattern between the study arms as reported by the OCT Corelab. The CoreLab will evaluate OCT images of each dissection including analysis of the length of the dissection, arc of the dissection, number of serrations, and the length of the serration.
Correlation of Luminal Gain and Plaque Modification | Baseline
  The correlation of the plaque modification achieved as determine from the OCT evaluation after treatment with the Study Device to the luminal gain achieved by conventional angioplasty as evaluated by the Core Lab.
Rate of Optimal PTA | Baseline
  Rate of procedures that achieve optimal PTA (<30% diameter stenosis without flow-limiting dissection measured by angiography)
Bail-out Stenting | Baseline
  Rate of bail-out stenting

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Columbia University, New York, New York
  - Weill Cornell Medical, New York, New York

IPD SHARING:
Plan to Share IPD: No